CLINICAL TRIAL: NCT00866112
Title: A Randomized Exercise Trial for Wheelchair Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Principal Investigator, Kathleen Grobe, Assitant Professor, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 10053
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2010-04

CONDITIONS: Spinal Cord Injury; Multiple Sclerosis; Muscular Dystrophy; Cerebral Palsy; Spina Bifida; Amputation; Arthritis; Stroke
Keywords: Wheelchair use; Spinal cord injury; Multiple sclerosis; Muscular dystrophy; Cerebral palsy; Spina bifida; Amputation; Arthritis; Stroke
MeSH Terms: conditions — Spinal Cord Injuries; Multiple Sclerosis; Muscular Dystrophies; Cerebral Palsy; Spinal Dysraphism; Arthritis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intervention group to promote physical activity
  Interventions: Other: Educational session to promote physical activity
- 2 (Other): Minimal contact control group
  Interventions: Other: Minimal contact

INTERVENTIONS:
Other: Educational session to promote physical activity — Educational session, goal setting, self monitoring of daily engagement in physical activity
  Arms: 1
Other: Minimal contact — Self guided education manual about adopting physical activity, self monitor daily engagement in physical activity
  Arms: 2

SUMMARY:
People with mobility disabilities are at greater risk than the general population for incurring health problems. Many of these conditions are preventable through behavior and lifestyle changes such as exercise and physical activity. Recent evidence suggests that people with disabilities experience the same physiologic response to exercise as the general population. Nonetheless, nearly three-fourths of those with disabilities report being entirely sedentary or not active enough to achieve health benefits. Despite some knowledge of issues that limit physical activity among this population, few studies have investigated methods for promoting physical activity adoption among people with disabilities, including wheelchair users. The purpose of this study is to test the effectiveness of a behavioral intervention to promote physical activity adoption over 6 months and maintenance of physical activity over another 6 months by community-dwelling manual wheelchair users.

ELIGIBILITY:
Inclusion Criteria:

* Be experiencing a permanent disability of at least 6 months that limits mobility sufficiently to require use of a wheelchair as the primary method of mobility outside the home
* Have not been moderately to vigorously physically active for the past 6 months
* Be willing to attend the educational workshop
* Receive physician approval for participation

Exclusion criteria include:

* Presence of medical conditions such as uncontrolled cardiovascular problems that the patient's physician identifies as being contraindicated for exercise
* Pregnancy or planning to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2008-05; Primary Completion 2011-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Weekly minutes spent in aerobic and strengthening activity | Baseline, 12, 26 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Froehlich-Grobe, PhD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas, Lawrence, Kansas, United States

REFERENCES:
- [Derived] Froehlich-Grobe K, Nary DE, VanSciver A, Washburn RA, Aaronson L. Truth be told: evidence of wheelchair users' accuracy in reporting their height and weight. Arch Phys Med Rehabil. 2012 Nov;93(11):2055-61. doi: 10.1016/j.apmr.2012.05.005. Epub 2012 May 15. PMID 22609118
- [Derived] Nary DE, Froehlich-Grobe K, Aaronson L. Recruitment issues in a randomized controlled exercise trial targeting wheelchair users. Contemp Clin Trials. 2011 Mar;32(2):188-95. doi: 10.1016/j.cct.2010.10.010. Epub 2010 Oct 27. PMID 21035565